CLINICAL TRIAL: NCT04156503
Title: A Pilot Study for the Quantitative Analysis of Positional Fatty Acids in Postprandial Chylomicron Triacylglycerol Using 13C NMR Spectroscopy
Brief Title: Pilot Study-Quantitative Analysis of Positional Fatty Acids in Postprandial Chylomicron Triacylglycerol Using 13C NMR Spectroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Malaysia Palm Oil Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PD222/17
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Chylomicron; fatty acid composition; lard; palm olein

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test fat: Palm olein (Experimental): One high fat muffin will be serves together with a glass of low fat milk shake.
  Interventions: Other: Palm olein vs Lard
- Test fat: Lard (Experimental): One high fat muffin will be serves together with a glass of low fat milk shake.
  Interventions: Other: Palm olein vs Lard

INTERVENTIONS:
Other: Palm olein vs Lard — A 5-hour postprandial feeding intervention with 2-weeks washout in between. Blood samples will be collected at hour 0 (baseline) before test meal, and hour 3, 4 and 5 after consumption of test meal.

SUMMARY:
13C NMR spectroscopy has been validated to be a rapid, direct and accurate quantitative method in determination of positional distribution of fatty acids in edible oils and fats, including the palm oil fractions (from soft olein to hard stearin). Nevertheless, there is paucity of literature describing its application in determining the positional fatty acid composition in blood triacylglycerols & biological samples, despite its widely used application in edible oils and fats. The postprandial feeding intervention is aimed to harvest chylomicron rich in triglycerides (~97% TAG) for NMR analysis.

DETAILED DESCRIPTION:
A pilot postprandial study with double blind, 2x2 arms randomized crossover experimental design will be carried out. A total of 10 subjects (5 males, 5 females) will be recruited and divided into 2 groups. Each group will be assigned to one of the test fat and fed with test meal prepared with 50g of test fats. 10 mL of blood samples will be collected at time points 0 (baseline, before meal) and 3, 4 and 5h after finish the meal. There shall be a 2-weeks washout period between each test fat.

Test fats used for this study are palm olein, with predominantly oleic acid at sn-2 position of the triglyceride backbone (about 68%, Gunstone et al, 2007) and lard, with predominantly palmitic acid at sn-2 position (about 72%, Gunstone et al., 2007). A high fat muffin with 50g of test fat will be formulated using the above two test fats mentioned. On each study day, a high fat muffin will be served and a glass of skim milk will be provided for subjects to help the digestion of fats from the muffins.

Chylomicron will be harvested using the ultracentrifugation technique. Samples collected will be stored in -80°C prior to NMR analysis.

ELIGIBILITY:
Inclusion Criteria:

* Non muslim, aged between 25 - 40 yrs old.
* BMI between 20 - 27.5 kg/m2.
* Blood pressure with <130mmHg for systolic pressure and < 80 mmHg for diastolic pressure.
* Blood glucose level in the range of 3.9 to 5.5 mmol/L.
* Total cholesterol level < 6.0 mmol/L.
* Triglycerides level < 2.3 mmol/L.
* No use of tobacco and no consumption of alcohol.

Exclusion Criteria:

* Suffer from chronic disease such as CVD, hypertension, diabetic, metabolic syndrome.
* Consuming any medical prescriptions/ supplements.
* Having blood clotting problem.
* Women who are pregnant or lactating.
* Hypertensive condition with systolic pressure >140mmHg and diastolic pressure > 90 mmHg.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Triglycerides profile in chylomicron harvested | Up to hour 5
  the positional composition of fatty acid in test fat that are retained upon absorption ( samples are pooled from 3, 4 &5 hour after test diet)

CONTACTS AND LOCATIONS:
Overall Officials: Phooi Tee Voon, Ph.D, Principal Investigator — MPOB
Locations (1):
- MalaysiaPOB, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No